CLINICAL TRIAL: NCT00242541
Title: Open Label Study Assessing the Efficacy and Safety of Octreotide Acetate in Patients With Acromegaly, With Micro or Macroadenomas
Brief Title: Study Assessing the Efficacy and Safety of Octreotide Acetate in Patients With Acromegaly, With Micro or Macroadenomas
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSMS995BMX02
Record Dates: First submitted 2005-10-09; First posted 2005-10-20 (Estimated); Last update posted 2012-04-26 (Estimated); Status verified 2012-04

CONDITIONS: Acromegaly
Keywords: microadenoma; macroadenoma
MeSH Terms: conditions — Acromegaly | interventions — Octreotide

ARMS (1):
- Octreotide acetate (Experimental)
  Interventions: Drug: Octreotide acetate

INTERVENTIONS:
Drug: Octreotide acetate
  Other Names: SMS995

SUMMARY:
The purpose of this study is to evaluate the efficacy of octreotide acetate to decrease GH and IGF-I levels in acromegalic patients, with microadenomas (≤ 10 mm) or macroadenomas (> 10 mm).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 - 80 years.
* Newly diagnosed or previously treated acromegalic patients.
* Lack of suppression of GH nadir to <1.0 microg/L, after oral administration of 75 g of glucose (OGTT).
* IGF-I levels above the upper limits of normal, i.e. 97th percentile (adjusted for age and gender).

Exclusion Criteria:

* Requires surgery for recent significant deterioration in visual fields or other neurological signs, which are related to the pituitary tumor mass.
* No evidence of pituitary adenoma on Magnetic Resonance Imaging (MRI).
* Symptomatic cholelithiasis.
* Unstable angina, sustained ventricular tachycardia, ventricular fibrillation, or a history of acute myocardial infarction within the three months preceding study entry.
* Liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis, or persistent ALT, AST, alkaline phosphatase 2 x > upper limit of normal, or total bilirubin 1.5 x > upper limit of normal.
* Female patients who are pregnant or lactating, or are of childbearing potential and not practicing a medically acceptable method for birth control. Medically acceptable methods include oral birth control pills, intrauterine devices, or mechanical methods (e.g. vaginal diaphragm, vaginal sponge or condom with spermicidal jelly). If oral contraception is used, the patient must have been practicing this method for at least two months prior to the screening visit and must agree to continue the oral contraceptive throughout the course of the study, and for one month after the study has ended.
* History of immunocompromise, including a positive HIV test result (ELISA and Western blot).

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2003-03; Primary Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the use of octreotide acetate to reduce levels of GH and IGF-I in Acromegalic patients with micro (< 10 mm) and macroadenomas (> 10 mm)

SECONDARY OUTCOMES:
Safety and tolerability of multiple doses
The efect of octreotide acetate in the tumor efect
To evaluate the capability to reduce sign and symptoms of Acromegaly

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Mexico City, Mexico